CLINICAL TRIAL: NCT05793918
Title: Percutaneous Electrolysis, Ultrasound-guided Percutaneous Neuromodulation Therapy and Eccentric Exercise in Supraspinatus Tendinopathy: A Single-Blind Randomized Controlled Trial.
Brief Title: Percutaneous Electrolysis, Ultrasound-guided Percutaneous Neuromodulation Therapy and Eccentric Exercise in Supraspinatus Tendinopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Percutaneous Electrolysis
Record Dates: First submitted 2023-03-15; First posted 2023-03-31 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-08

CONDITIONS: Supraspinatus Tendinitis
Keywords: tendinopathy; electrolysis; exercise; dry needling
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the supraspinatus tendinopathy.
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Electrolysis and neuromodulation. (Experimental): The intervention for this group consisted of Therapeutic Percutaneous Electrolysis and neuromodulation. Patient received once week for four weeks associated with eccentric exercises device at home.
  Interventions: Other: Therapeutic Percutaneous Electrolysis an neuromodulation
- Control group (Active Comparator): The multimodal physical therapy program includes 10 sessions of:
  Ultrasound pulsatil therapy (US) for 10 minutes , transcutaneous electric nerve stimulation (TENS) for 20 minutes ans associated with eccentric exercises device at home.
  Interventions: Other: Conventional group

INTERVENTIONS:
Other: Therapeutic Percutaneous Electrolysis an neuromodulation — Therapeutic Percutaneous Electrolysis an neuromodulation associated with eccentric exercises devices at home.
  Arms: Percutaneous Electrolysis and neuromodulation.
Other: Conventional group — Ultrasound pulsatil therapy (US), transcutaneous electric nerve stimulation (TENS) for 20 minutes and associated with eccentric exercises devices at home.
  Arms: Control group

SUMMARY:
The supraspinatus muscle tendinopathy show a big impact, however, there is a lack of awareness about the options of the physiotherapist treatment. It is necessary to do studies about effectiveness of therapeutic percutaneous electrolysis and neuromodulation. This technique enables treatment of the tendinopathies. To analyze the effectiveness of therapeutic percutaneou electrolysis and neuromodulation in the treatment of supraspinatus muscle tendinopathy. Single center randomized controlled trial, parallel treatment design. A specialist physician will be diagnosed the supraspinatus muscle tendinopathy. Participants will be randomly assigned to receive treatmen for 4 weeks: percutaneou electrolysis and neuromodulation associated with eccentric exercises or conventional treatment of Physiotherapy with the same eccentric exercises. Both interventions were performed under ultrasound guidance with a portable ultrasound (General Electric LogicE). Data will be collected by a blinded evaluator.

DETAILED DESCRIPTION:
Eccentric exercises of the supraspinatus muscle were performed in 3 sets of 10 repetitions. Participants were asked to perform the exercise program on an individual basis twice every day for 4 weeks. The eccentric program consisted of 3 exercises, focusing on the supraspinatus, infraspinatus, and scapular muscles. Participants were asked to do a normal abduction (concentric phase) and a slow return to the initial position (eccentric phase) included first the concentric phase, and the eccentric phase was slowly conducted. The exercise program was taught by a physiotherapist in the first session and monitored in the subsequent sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with supraspinatus tendinopathies that do not improve with conventional physiotherapy or pharmacological therapy protocols.
* Subjects who are in an active state of pain, who present painful symptoms in a sensitive and painful area of the tendon of insertion of the supraspinatus muscle in the humerus.

Exclusion Criteria:

* Individuals who have received surgery intervention in the same shoulder, or have suffered fractures or dislocations in the same shoulder.
* Individuals have received the proposed treatment in one month´s period previously.
* Individuals who suffering from cervical radiculopathies, fibromialgia síndrome, cardiac patients with pacemakers, cancer, infectious processes, or generalized lymphedema.
* Pregnant women can not receive this treatment intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
The intensity of shoulder pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).

SECONDARY OUTCOMES:
The intensity of shoulder pain. | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
The intensity of shoulder pain | Twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
Questionnaire DASH. | Baseline, four, twelve weeks and twenty four weeks.
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-re, four, twelve weeks and twenty four weeks.
Scale SPADI. | Baseline, four, twelve weeks and twenty four weeks.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. Both dimensions account for 50% of the overall score, and scores from 0 to 100.
Active shoulder range of motion | Baseline, four, twelve weeks and twenty four weeks.
  The range of motion will be evaluated in flexion, extension, internal rotation, external rotation and abduction with a goniometric
Pressure pain thresholds in supraspinatus trigger points | Baseline, four, twelve weeks and twenty four weeks.
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline, Pain TestTM, Wagner Instruments). The clinimetric properties of this instrument have been evaluated previously. The PPT will the point at which pressure elicited pain and will presented as kilograms per square centimeter. All measurements will be conducted by the same well-trained physician.
Questionnaire SF 12 | Baseline, four, twelve weeks and twenty four weeks.
  SF-12 questionnaire is a reliable measure of perceived health that describes the degree of general physical health status and mental health distress. It consists of 12 items, derived from the physical and mental domains. In our study SF-12 was considered altered if the score was <40, either from the physical or mental functioning point of view, because means of 50 and standard deviations of 10 are usually achieved in the general population.
GROCS scale | Baseline, four, twelve weeks and twenty four weeks.
  The multidimensional health related quality of life.
The jobe test | Baseline, four, twelve weeks and twenty four weeks.
  Jobe's test assesses for possible supraspinatus weakness and/or impingement.
The Neer test | Baseline, four, twelve weeks and twenty four weeks.
  The Neer test is performed to check for compression of the rotator cuff tendons at the coracoacromial arch.
Hawkins-Kennedy test | Baseline, four, twelve weeks and twenty four weeks.
  the Hawkins-Kennedy test is a test for impingement in the shoulder

CONTACTS AND LOCATIONS:
Overall Officials: manuel rodriguez huguet, Physiotherapy, Study Director — University of Cádiz
Locations (1):
- Policlínica Santa María, Cadiz, Cádiz, Spain

REFERENCES:
- [Background] Cook JL, Purdam CR. Is tendon pathology a continuum? A pathology model to explain the clinical presentation of load-induced tendinopathy. Br J Sports Med. 2009 Jun;43(6):409-16. doi: 10.1136/bjsm.2008.051193. Epub 2008 Sep 23. PMID 18812414
- [Background] McCreesh K, Lewis J. Continuum model of tendon pathology - where are we now? Int J Exp Pathol. 2013 Aug;94(4):242-7. doi: 10.1111/iep.12029. PMID 23837792
- [Background] Khan KM, Cook JL, Maffulli N, Kannus P. Where is the pain coming from in tendinopathy? It may be biochemical, not only structural, in origin. Br J Sports Med. 2000 Apr;34(2):81-3. doi: 10.1136/bjsm.34.2.81. No abstract available. PMID 10786860
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Rodriguez-Huguet P, Ibanez-Vera AJ, Rodriguez-Almagro D, Martin-Valero R, Diaz-Fernandez A, Lomas-Vega R. Effectiveness of Percutaneous Electrolysis in Supraspinatus Tendinopathy: A Single-Blinded Randomized Controlled Trial. J Clin Med. 2020 Jun 12;9(6):1837. doi: 10.3390/jcm9061837. PMID 32545583
- [Background] Lewis JS. Rotator cuff tendinopathy. Br J Sports Med. 2009 Apr;43(4):236-41. doi: 10.1136/bjsm.2008.052175. Epub 2008 Sep 18. PMID 18801774
- [Background] Osborne JD, Gowda AL, Wiater B, Wiater JM. Rotator cuff rehabilitation: current theories and practice. Phys Sportsmed. 2016;44(1):85-92. doi: 10.1080/00913847.2016.1108883. Epub 2015 Nov 7. PMID 26548634
- [Background] Garcia Bermejo P, De La Cruz Torres B, Naranjo Orellana J, Albornoz Cabello M. Autonomic Responses to Ultrasound-Guided Percutaneous Needle Electrolysis: Effect of Needle Puncture or Electrical Current? J Altern Complement Med. 2018 Jan;24(1):69-75. doi: 10.1089/acm.2016.0339. Epub 2017 Jan 30. PMID 28135129
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Lomas-Vega R, Martin-Valero R, Diaz-Fernandez A, Obrero-Gaitan E, Ibanez-Vera AJ, Rodriguez-Almagro D. Percutaneous Electrolysis in the Treatment of Lateral Epicondylalgia: A Single-Blind Randomized Controlled Trial. J Clin Med. 2020 Jul 1;9(7):2068. doi: 10.3390/jcm9072068. PMID 32630241
- [Background] Littlewood C, Ashton J, Chance-Larsen K, May S, Sturrock B. Exercise for rotator cuff tendinopathy: a systematic review. Physiotherapy. 2012 Jun;98(2):101-9. doi: 10.1016/j.physio.2011.08.002. Epub 2011 Oct 5. PMID 22507359
- [Background] Dejaco B, Habets B, van Loon C, van Grinsven S, van Cingel R. Eccentric versus conventional exercise therapy in patients with rotator cuff tendinopathy: a randomized, single blinded, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):2051-2059. doi: 10.1007/s00167-016-4223-x. Epub 2016 Jun 28. PMID 27351548
- [Background] Heron SR, Woby SR, Thompson DP. Comparison of three types of exercise in the treatment of rotator cuff tendinopathy/shoulder impingement syndrome: A randomized controlled trial. Physiotherapy. 2017 Jun;103(2):167-173. doi: 10.1016/j.physio.2016.09.001. Epub 2016 Sep 21. PMID 27884499
- [Background] Kinsella R, Cowan SM, Watson L, Pizzari T. A comparison of isometric, isotonic concentric and isotonic eccentric exercises in the physiotherapy management of subacromial pain syndrome/rotator cuff tendinopathy: study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2017 Nov 14;3:45. doi: 10.1186/s40814-017-0190-3. eCollection 2017. PMID 29163981
- [Background] Lin ML, Chiu HW, Shih ZM, Lee PY, Li PZ, Guo CH, Luo YJ, Lin SC, Lin KY, Hsu YM, Pang A, Pang W. Two Transcutaneous Stimulation Techniques in Shoulder Pain: Transcutaneous Pulsed Radiofrequency (TPRF) versus Transcutaneous Electrical Nerve Stimulation (TENS): A Comparative Pilot Study. Pain Res Manag. 2019 Feb 4;2019:2823401. doi: 10.1155/2019/2823401. eCollection 2019. PMID 30863472